CLINICAL TRIAL: NCT06378346
Title: GU-01: Glycyrrhizin in Prostate Cancer: A Window-of-Opportunity Trial
Brief Title: GU-01: Glycyrrhizin in Prostate Cancer
Acronym: GU-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Natalie Reizine, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-077
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation; Glycyrrhizic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Observational Arm 1 (Dose Level 0) (Placebo Comparator): 10 participants will be randomized to observational arm
  Interventions: Other: Observation
- Glycyrrhizin Arm 2 (Dose Level 1) (Experimental): 25 participants will be randomized to receive 75mg daily for 6 weeks (+/- 2 weeks)
  Interventions: Drug: Glycyrrhizin - 75 mg
- Glycyrrhizin Arm 3 (Dose Level 2) (Experimental): 25 participants will be randomized to receive 150mg daily for 6 weeks (+/- 2 weeks)
  Interventions: Drug: Glycyrrhizin - 150 mg

INTERVENTIONS:
Other: Observation — Participants will not receive glycyrrhizin
  Arms: Observational Arm 1 (Dose Level 0)
Drug: Glycyrrhizin - 75 mg — Participants will either receive 75 mg orally daily
  Arms: Glycyrrhizin Arm 2 (Dose Level 1)
Drug: Glycyrrhizin - 150 mg — Participants will receive 150 mg orally daily
  Arms: Glycyrrhizin Arm 3 (Dose Level 2)

SUMMARY:
This is a pilot, randomized, window-of-opportunity treatment trial in which participants with previously untreated prostate cancer (PCa) who are candidates for surgery (radical prostatectomy)

DETAILED DESCRIPTION:
This is a pilot, randomized, window-of-opportunity treatment trial in which participants with previously untreated prostate cancer who are candidates for surgery (radical prostatectomy) will receive one cycle of therapy consisting of Glycyrrhizin (GLY) (Observation, Dose Level 1 75mg daily, or Dose Level 2, 150mg daily) for 6 weeks (+/- 2 weeks) prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at time of consent
2. ECOG performance status of 0, 1, or 2
3. Histologic diagnosis of prostate cancer
4. Patient suitable for radical prostatectomy as determined by surgical team
5. Able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
6. Willing to use barrier contraceptive method during study intervention

Exclusion Criteria:

1. Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating urologic oncology team.
2. Previous chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents and/or investigational agents within 30 days of starting study treatment.
3. Potent or moderate inhibitors and inducers of CYP3A4 if taken within a 1 week wash-out period
4. Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation, or History of Torsades de Pointes. This may include patients who have sub-optimally controlled hypertension, serum potassium levels <4.0 mEq/L, serum magnesium ≤1.8 mg/dL, prolonged gastrointestinal transit time, or decreased 11-β-hydroxysteriod dehydrogenase-2 activity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate anti-tumor activity of GLY by assessing changes in prostate-specific antigen (PSA) after GLY treatment administration and prior to radical prostatectomy | 2 months
  Changes in prostate specific antigen (PSA) in patients with prostate cancer will be assessed before and after administration of GLY

SECONDARY OUTCOMES:
To evaluate the tolerability of GLY treatment administered daily prior to prostatectomy. | 2 months
  Tolerability will be assessed by NCI Common Terminology Criteria for Adverse Events (AE) (NCI CTCAE) Version 5 (v5.0). The safety rate is calculated as the proportion of patients without Grade 2 or higher AE.
To assess of clinical laboratory and pathologic correlates in patients in relation to GLY treatment administration | 2 months
  Clinical laboratory and pathologic correlates that will be assessed include:
  * Plasma GLY levels,
  * Blood chemistries (sodium, potassium, serum creatinine or eGFR),
  * Fasting serum glucose, insulin, and lipid levels,
  * Serum testosterone and dehydroepiandrosterone sulfate (DHEA-S) levels,
  * Inflammatory markers (C-Reactive Protein, interleukin-1β, Tumor necrosis factor α, and interleukin-1β),
  * Serum levels of growth factors (vascular endothelial growth factor, hepatocyte growth factor, Insulin-like growth factor-1, and insulin-like growth factor binding protein-3),
  * Gene expression analysis evaluating prostate tumor signaling pathways
  * Ki67, SOX2, and AR expression in tumor specimens obtained before and after administration of GLY as assessed by IHC, and
  * The concentration of GLY in tumor specimens
To evaluate patient perspectives on clinical trial enrollment and complementary and integrative medicine (CAM) approaches as evaluated through survey questionnaires | 2 months
  Surveys will be administered before and after GLY treatment

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Reizine, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States